CLINICAL TRIAL: NCT06688292
Title: A Randomized, Safety and Efficacy Study of Taneasy 600mg Granules and Actein Effervescent Tablets 600MG in COPD Subjects
Brief Title: The Safety and Effectiveness of Taneasy and Actein in COPD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bun Yao Biotechnology Co., Ltd (Industry)
Collaborators: KGS Pharmamate Co., Ltd (Unknown); Taichung Veterans General Hospital, Taichung (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCQ230209TC
Record Dates: First submitted 2024-11-11; First posted 2024-11-14 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-12

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Taneasy 600mg granules (Experimental): Dose： 600 mg/time. Use ：two times per day.
  Interventions: Drug: Taneasy 600mg granules
- Actein effervescent tablets 600MG (Active Comparator): Dose： 600 mg/time. Use ：two times per day
  Interventions: Drug: Actein effervescent 600mg

INTERVENTIONS:
Drug: Taneasy 600mg granules — Treatment of respiratory affections characterized by thick and viscous hypersecretion due to acute bronchitis,chronic bronchitis and its exacerbation, plumonary emphysema,mucoviscidosis and bronchiectasis.
  Arms: Taneasy 600mg granules
Drug: Actein effervescent 600mg — Treatment of respiratory affections characterized by thick and viscous hypersecretion due to acute bronchitis,chronic bronchitis and its exacerbation, pulmonary emphysema, mucoviscidosis and bronchiectasis.
  Other Names: acetylcysteine effervesecent 600mg
  Arms: Actein effervescent tablets 600MG

SUMMARY:
To evaluate the safety and efficacy of Taneasy 600mg granules and Actein effervescent tablets 600MG administered twice daily for 14 days in treatment of COPD Disease.

DETAILED DESCRIPTION:
The study will enroll 40~60 patients and complete 40 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged older than 20~75 years old.
2. Able to sign informed consent prior to the study.
3. Subjects have COPD.

Exclusion Criteria:

1. Subjects with known hypersensitivity to Acetylcysteine preparations.
2. Subjects with other serious medical diseases that are judged by the attending physician to affect the evaluation results (such as: tuberculosis, pneumonia, bronchial asthma, bronchiectasis, cor pulmonale, lung cancer, acute myocardial infarction, acute hepatitis, renal failure, etc.)
3. Pregnancy or breast-feeding woman.
4. Female subjects or their sexual partners do not use contraception during the trial.
5. Joining any drug clinical trial within 3 months prior to dosing.
6. Investigator considered to be inappropriate for enrollment.
7. Phenylketonuria (PKU).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2024-09-20 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of Taneasy 600mg granules and Actein effervescent tablets 600MG administered twice daily for 14 days in treatment of COPD Disease. | one month
  Primary Evaluation Criteria:
  CAT score (COPD Assessment Test) The maximum score is 40. Higher scores indicate your COPD has a greater impact on your overall health and well-being.

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No